CLINICAL TRIAL: NCT05930392
Title: Comparative Evaluation of Microsurgery vs Conventional Surgical Technique of Gingival Depigmentation on Pink Esthetics and Patient-related Outcomes: A Split-mouth Randomised Controlled Clinical Study.
Brief Title: Comparative Evaluation of Microsurgery vs Conventional Surgical Technique of Gingival Depigmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AANCHALSAHNIPERIO2
Record Dates: First submitted 2023-05-04; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Gingival Pigmentation; Melanosis
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GINGIVAL DEPIGMENTATION USING MICROSURGERY (Active Comparator): Surgical excision of hyper-pigmented gingival tissue using microsurgical blade (keratome 2.2) and magnification loupes under local anaesthesia. Application of periodontal dressing followed by post-operative instructions.
  Interventions: Procedure: Gingival depigmentation using microsurgery
- Conventional surgical technique of gingival depigmentation (Active Comparator): Surgical excision of hyper-pigmented gingival tissue using conventional surgical blade (#15) under local anaesthesia. Application of periodontal dressing followed by post-operative instructions.
  Interventions: Procedure: Conventional surgical depigmentation

INTERVENTIONS:
Procedure: Gingival depigmentation using microsurgery — GINGIVAL DEPIGMENTATION USING MICROSURGICAL BLADE AND MAGNIFICATION LOUPES
  Arms: GINGIVAL DEPIGMENTATION USING MICROSURGERY
Procedure: Conventional surgical depigmentation — GINGIVAL DEPIGMENTATION USING CONVENTIONAL SURGICAL TECHNIQUE
  Arms: Conventional surgical technique of gingival depigmentation

SUMMARY:
Gingiva being the most frequently pigmented tissue of the oral cavity challenges a lot of people with an esthetic concern. Increased production of melanin, a pigment produced by the melanocytes present in the basal and suprabasal cell layers of the epithelium leads to the hyper-pigmented appearance. Over the decades many non-surgical as well as surgical techniques have been developed to manage the melanin induced hyper-pigmentation of gingival tissue with comparable efficacies. Till date, the most common gingival depigmentation procedure with satisfactory results remains the conventional scalpel (#15 blade) method. Nowadays, minimally traumatising the surgical field and gaining maximum outputs with help of microscopy and microsurgical instruments has attained a level of utmost importance in surgical procedures including periodontal therapy. Improved results in terms of increased vascularization of the grafts, relatively better percentages of root coverage a significant increase in width and thickness of keratinized tissue, an improved esthetic outcome and decreased patient morbidity in cases of gingival recession treated via microsurgical approach have been observed and well documented. However, perusal of the literature available suggests that clinical outcomes and esthetic potential of the results of gingival depigmentation using principles of microsurgery is an area of interest that still needs to be explored further. This study is therefore aimed at evaluating and comparing the clinical, esthetic and patient-related outcomes of gingival depigmentation performed using microsurgery vs conventional surgical technique.

DETAILED DESCRIPTION:
AIM: To evaluate and compare the clinical, esthetic and patient-related outcomes of gingival depigmentation performed via microsurgery vs conventional surgical technique.

OBJECTIVES:

1. To evaluate and compare melanin pigmentation using Dummett Oral Pigmentation Index (DOPI), Hedin melanin index (HMI) between both the treatment modalities at baseline, 1 week, 1 month and 3 months post-operatively.
2. To assess a) patient-related outcome measures (PROMs) such as post-operative pain perception/discomfort on a visual analog scale (VAS) , patient's preference of the mode of treatment /esthetic satisfaction and b) clinical parameters such as bleeding, redness, swelling, wound healing, gingival colour, gingival morphology at baseline, within 24 hours, 1 week, 1 month and 3 months.
3. To evaluate the effect of different treatment modalities on melanocyte histopathologic count (MHC).

TIME FRAME: 3 months SAMPLE SIZE: To achieve a power of 80%, level of significance of 5% and assuming an effect size of 0.8, a minimum sample size of 18 patients is needed in each group. Accounting for a 20% drop out rate, 22 patients are needed in each group.

METHODOLOGY: Patients fulfilling the eligibility criteria will be enrolled in the study after obtaining an informed written consent. A split-mouth design with maxillary and mandibular anteriors being randomly allocated into test (microsurgery) and control (conventional surgical depigmentation) technique to each patient using a radio-opaque box having 44 chits.

STATISTICAL ANALYSIS: Data recorded will be processed by standard statistical analysis. The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. If it is in normal distribution, intra group comparison will be done by paired t-test between two time points and inter group comparison will be done by using unpaired t-test between two groups. If it is in non-normal distribution, intra group comparison will be done by Wilcoxon signed rank test and inter group comparison will be done by Mann-Whitney U test.

SETTING: Department of Periodontology and Oral Implantology, PGIDS, Rohtak, Haryana.

STUDY DESIGN: Split-mouth Comparative Randomised Controlled Clinical Study.

ELIGIBILITY:
Inclusion Criteria:

1)Systemically healthy patients seeking treatment for gingival hyper-pigmentation

Exclusion Criteria:

1. Gingival index (Loe and Sillness 1963) of greater than or equal to 1 at any site of surgical field.
2. patients with periodontitis
3. patients with pathologic or drug-induced gingival hyper-pigmentation
4. patients with history of systemic illness with the potential to influence the periodontal status or outcome of periodontal intervention;
5. patients with Miller Grade II /Grade III tooth mobility;
6. patients taking medications such as NSAIDS, corticosteroids, statins or calcium channel blockers, which are known to influence periodontal status;
7. pregnant or lactating women;
8. history of use of tobacco;

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
CLINICAL PARAMETER- Bleeding | 3 MONTHS
  bleeding score classified in accordance to Ishi et al and Kawashima et al
  A: NONE B: SLIGHT C: MODERATE D: SEVERE
CLINICAL PARAMETER- REDNESS | 3 MONTHS
  redness score classified in accordance to Ishi et al and Kawashima et al
  A: NONE B: SLIGHT C: MODERATE D: SEVERE
CLINICAL PARAMETER- swelling | 3 MONTHS
  swelling score classified in accordance to Ishi et al and Kawashima et al
  A: NONE B: SLIGHT C: MODERATE D: SEVERE
CLINICAL PARAMETER- WOUND HEALING | 3 MONTHS
  Wound healing score classified in accordance to Ishi et al and Kawashima et al
  A: COMPLETE EPITHELIALIZATION B: INCOMPLETE OR PARTIAL EPITHELIALIZATION C: ULCER D: TISSUE DEFECT OR NECROSIS
CLINICAL PARAMETER- Gingival color | 3 MONTHS
  Gingival Color
  A: IMPROVEMENT B: SLIGHT IMPROVEMENT C: NO CHANGE D: DETERIORATION
DUMMETT ORAL PIGMENTATION INDEX (DOPI) | 3 MONTHS
  DOPI
  Score Criteria 0 Pink tissue (no clinical pigmentation)
  1. Mild light brown tissue (mild clinical pigmentation)
  2. Medium brown or mixed brown and pink tissue (moderate clinical pigmentation)
  3. Deep brown/ blue-black tissue (heavy clinical pigmentation)
HEDIN MELANIN INDEX (HMI) | 3 MONTHS
  HMI
  Score Criteria 0 No pigmentation
  1. One or two solitary units of pigmentation in the papillary gingiva
  2. >3 units of pigmen- tation in the papillary gingiva without formation of a continuous ribbon
  3. More than equal to 1 short continuous ribbons of pigmentation
  4. One continuous ribbon including the entire area between the canines
Patient-related outcome measures (PROMs) - post-operative pain perception | 3 months
  Pain will be assessed on a 100-mm horizontal, continuous interval scale with the left endpoint marked ''no pain'' and the right endpoint marked ''worst pain.'' The patient placed a mark to coincide with the level of pain. Scores were calculated as: 0 = no pain; 0.1 to 3.0 cm (1 to 30 mm) = slight pain; 3.1 to 6.0 cm (31 to 60 mm) = moderate pain; 6.1 to 10 cm (61 to 100 mm) = severe pain.
Patient-related outcome measures (PROMs) - ESTHETIC SATISFACTION | 3 months
  ESTHETIC SATISFACTION WILL BVE EVALUATED AS PER PATIENT'S RESPONSE TO PREFERRED CHOICE OF TREATMENT - CONVENTIONAL OR MICROSURGICAL

SECONDARY OUTCOMES:
MELANOCYTE HISTOPATHOLOGIC COUNT (MHC) | 3 MONTHS
  EFFECT ON MELANOCYTE HISTOPATHOLOGIC COUNT
  The activity of the melanocytes will be measured at baseline and 3 months post-operatively, by microscopically viewing the density of melanin granules.35 The grading will be done using the following scale: 0 = absence of melanin granules (no pigmentation); 1 = rare and scattered melanin granules (mild pigmentation); 2 = dense but not aggregated melanin granules (moderate pigmentation); or 3 = dense and aggregated melanin granules (heavy pigmentation).
PERIODONTAL PARAMETER - PLAQUE INDEX | 3 MONTHS
  PLAQUE INDEX
  " SCORE" "CRITERIA" 0 No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque could only be recognized by running a probe across the tooth surface area
  2. Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin, which can be seen with the naked eyes.
  3. Abundance of soft matter on tooth and/or on the gingival margin.
PERIODONTAL PARAMETERS - GINGIVAL INDEX, | 3 MONTHS
  GINGIVAL INDEX
  Score Criteria 0 Absence of inflammation/normal gingiva.
  1. Mild inflammation, slight change in colour, slight oedema; no bleeding on probing within 30 seconds.
  2. Moderate inflammation; moderate glazing, redness, oedema, hypertrophy and bleeding on probing.
  3. Severe inflammation; marked redness and hypertrophy ulceration of gingival margin. Tendency to spontaneous bleeding.
PERIODONTAL PARAMETERS - BLEEDING ON PROBING (BOP) | 3 MONTHS
  BLEEDING ON PROBING
  BOP will be recorded as 1 (present) if it occurs within 15 secs of probing and 0 (absent) if no bleeding occurs. It will be calculated in %. After adding all the scores, total score will be divided by the total number of surfaces accessed and multiplied by 100. It will be designed as % sites
PERIODONTAL PARAMETER - PROBING POCKET DEPTH (PPD) | 3 MONTHS
  PROBING POCKET DEPTH
  Probing pocket depth will be measured as the distance from the gingival margin to the base of pocket. The probing depth measurements will be assessed using a calibrated manual periodontal probe (PCP-UNC 15 Hu-Friedy, Chicago, IL, USA). The probe will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of each tooth - mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual. Measurements will be rounded to the nearest whole millimetre.
PERIODONTAL PARAMETER - CLINICAL ATTACHMENT LEVEL (CAL) | 3 MONTHS
  CLINICAL ATTACHMENT LEVEL Clinical Attachment Level will be measured as the distance between the base of the pocket and the cemento-enamel junction (CEJ). Measurements will be made at 6 sites of each tooth- mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual using UNC-15 probe.
PERIODONTAL PARAMETERS - GINGIVAL RECESSION (GR) | 3 MONTHS
  GINGIVAL RECESSION
  Recession will be measured as the vertical distance from the CEJ to the deepest part of gingival margin in the middle of the buccal aspect of the crown.

CONTACTS AND LOCATIONS:
Overall Officials: AANCHAL SAHNI, BDS, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES,ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India